CLINICAL TRIAL: NCT05476328
Title: A Feasibility, Prospective, Repeated-measures Investigation to Investigate Innovations in Sound Processing in Adult and Paediatric Recipients Implanted With CE Approved Nucleus Cochlear Implants: an Umbrella Investigation.
Brief Title: Sound Processing Innovations in Adult and Paediatric Cochlear Implant Recipients.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cochlear (Industry)
Collaborators: Trium Clinical Consulting (Industry); Avania (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: AI5762
Record Dates: First submitted 2022-06-27; First posted 2022-07-27 (Actual); Results first posted 2025-02-13 (Actual); Last update posted 2025-02-13 (Actual); Status verified 2025-02

CONDITIONS: Hearing Loss
MeSH Terms: conditions — Hearing Loss | interventions — Equipment and Supplies

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- All Participants (Other): Advanced Combination Encoder (ACE) sound processing strategy (reference strategy), Spread Precompensation Advanced Combination Encoder (SPACE), and Optimised Pitch and Language strategy-SPACE (OPAL-SPACE; combined OPAL and SPACE strategy) were evaluated in adult cochlear implant recipients. The evaluation order of sound strategies was counterbalanced. All strategies were programmed using a research version of Custom Sound and the investigational software: Cochlear Device Interface Tool (CDI Tool).
  Interventions: Device: SPACE; Device: OPAL-SPACE; Device: ACE; Device: Cochlear Device Interface (CDI) Tool

INTERVENTIONS:
Device: SPACE — SPACE (Spread Precompensation Advanced Combination Encoder) is a sound coding strategy that is intended to improve spectral resolution, and hence hypothesised to improve cochlear implant (CI) speech understanding in noise. It is an alternative to the ACE sound coding strategy. It has been implemented on the Nucleus 7 CP1000 sound processor for CIC4-based implants.
  Other Names: Spread Precompensation Advanced Combination Encoder
Device: OPAL-SPACE — OPAL-SPACE (combined OPAL and SPACE strategy) aims to preserve as many of the significant features encoded by both OPAL and SPACE strategies individually. Since SPACE codes spectral envelope information, while OPAL codes temporal periodicity information, it is reasonable to suggest that both coding techniques can be combined to improve perception additively.
Device: ACE — Advanced Combination Encoder (ACE) is the commercially available, reference sound processing strategy.
  Other Names: Advanced Combination Encoder
Device: Cochlear Device Interface (CDI) Tool — For all strategies, programming will be performed using a research version of Custom Sound and the investigational software: Cochlear Device Interface Tool (CDI Tool). Investigational software will be used to stream stimulation sequences to a commercially available N6 sound processor using the Cochlear NIC4.1 interface.

SUMMARY:
This is a feasibility, prospective with sequential enrolment, multicenter, clinical investigation in adults and paediatrics with a CE approved Nucleus cochlear implant.

Subjects older than 5 years will be included. Subjects will be screened and up to 120 eligible subjects will be recruited in the clinical investigation.

Subjects will attend scheduled study visits over a period up to 5 years in different sub-studies as described in the sub-study documentation.

A clinical setting can consist of therapeutic elements and evaluations. Subjects will be assessed with the commercially available Nucleus sound processor or via the xPC, NIC, etc. if required. Acute testing will be done where possible. Take home use will be applied when learning effects may play a significant role and to evaluate the acceptance of the new or improved sound coding algorithm or signal processing, in as many listening environments as possible. The subject might also be asked to complete questionnaires, to perform at-home tests etc. during this take home use and/or at the clinical visits. The time for a clinical visit will be limited to a maximum of 4 hours. The time in between clinical visits will vary with typical spacing of between 0 (acute) to 4 weeks.

The goals of this umbrella investigation are to measure hearing outcomes to assess performance and/or to achieve higher convenience for implant users and hearing care professionals. The outcomes of the study will guide Cochlear to select features for inclusion in future Nucleus cochlear implant systems and/or future models of care.

ELIGIBILITY:
Inclusion Criteria:

* Users of a CE approved Nucleus cochlear implant, resulting in open set speech understanding.
* Paediatrics: Older than 5 years and <18 years when entering the study. (Belgium only) or
* Adults: ≥18 years when entering the study (Belgium and Australia).
* Subject/legally designated representative is fluent speaker in the language used for assessments.
* Willing and able to provide written informed consent (for paediatric populations this criterion applies to the parent/ legally designated representative).

Exclusion Criteria:

* Unable or unwilling to comply with the requirements of the clinical investigation as determined by the investigator.
* Additional health factors, known to the investigator, that would prevent or restrict participation in the audiological evaluations.
* Investigator site personnel directly affiliated with this study and/or their immediate families; immediate family is defined as a spouse, parent, child, or sibling.
* Cochlear employees or employees of Contract Research Organisations or contractors engaged by Cochlear for the purposes of this investigation.
* Currently participating, or participated within the last 30 days, in another interventional clinical investigation/trial involving an investigational drug or device.

Min Age: 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2020-01-22 (Actual); Primary Completion 2023-03-17 (Actual); Study Completion 2023-03-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Komal Arora, Study Director — Cochlear
Locations (5):
- Australia (2):
  - HEARnet Clinical Studies, Carlton, Victoria
  - Cochlear Ltd. Melbourne, East Melbourne
- Belgium (3):
  - AZ Sint-Jan Brugge-Oostende AV, Bruges
  - Cochlear Technology Centre Belgium, Mechelen
  - Sint-Augustinus Antwerpen, Wilrijk

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The participant flow includes only one group as this was a repeated measures, single-arm study where all participants were exposed to all sound processing strategies. Data from the same participants was collected multiple times across different conditions. The focus was on assessing effects within the same group under varying conditions, making it a single-arm design with repeated measurements on each participant.
Groups:
- All Participants: Advanced Combination Encoder (ACE) sound processing strategy (reference strategy), Spread Precompensation Advanced Combination Encoder (SPACE), and Optimised Pitch and Language strategy-SPACE (OPAL-SPACE; combined OPAL and SPACE strategy) were evaluated in adult cochlear implant recipients. All strategies were programmed using a research version of Custom Sound and the investigational software: Cochlear Device Interface Tool (CDI Tool).
  SPACE: SPACE (Spread Precompensation Advanced Combination Encoder) is a sound coding strategy that is intended to improve spectral resolution, and hence hypothesised to improve cochlear implant (CI) speech understanding in noise. It is an alternative to the ACE sound coding strategy. It has been implemented on the Nucleus 7 CP1000 sound processor for CIC4-based implants.
  OPAL-SPACE: OPAL-SPACE (combined OPAL and SPACE strategy) aims to preserve as many of the significant features encoded by both OPAL and SPACE strategies individually. Since SPACE codes spectral envelope information, while OPAL codes temporal periodicity information, it is reasonable to suggest that both coding techniques can be combined to improve perception additively.
  ACE: Advanced Combination Encoder (ACE) is the commercially available, reference sound processing strategy.
  Cochlear Device Interface (CDI) Tool: For all strategies, programming will be performed using a research version of Custom Sound and the investigational software: CDI Tool.
Period: Overall Study
Arm/Group | All Participants
Started | 8
ACE Strategy | 8
SPACE Strategy | 8
OPAL-SPACE Strategy | 8
Completed | 8
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | All Participants
Number analyzed (Participants) | 8
Age, Continuous [Mean (Full Range); unit: years] | 69 [61 to 76]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 5
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Clinical Device in Test Ear [Count of Participants; unit: Participants]
  N7 CI24RE | 3
  N7 CI512 | 5

OUTCOME MEASURES:

1. Primary Outcome: Monosyllabic Word in Quiet Scores.
Description: Monosyllabic word in quiet scores (for conventional Advanced Combination Encoders and new sound coding strategy). Resultant score is percentage of words repeated correctly. Possible scores ranges from 0% to 100% correctly repeated. Higher percentage score means better outcome
Time Frame: One Day
Measure: Mean (Standard Deviation); unit: Percentage of words repeated correctly
Groups:
- All Participants: Advanced Combination Encoder (ACE) sound processing strategy (reference strategy), Spread Precompensation Advanced Combination Encoder (SPACE), and Optimised Pitch and Language strategy-SPACE (OPAL-SPACE; combined OPAL and SPACE strategy) were evaluated in adult cochlear implant recipients. All strategies were programmed using a research version of Custom Sound and the investigational software: Cochlear Device Interface Tool (CDI Tool).
  SPACE is a sound coding strategy that is intended to improve spectral resolution, and hence hypothesised to improve cochlear implant (CI) speech understanding in noise. It is an alternative to the ACE sound coding strategy. It has been implemented on the Nucleus 7 CP1000 sound processor for CIC4-based implants.
  OPAL-SPACE aims to preserve as many of the significant features encoded by both OPAL and SPACE strategies individually. Since SPACE codes spectral envelope information, while OPAL codes temporal periodicity information, it is reasonable to suggest that both coding techniques can be combined to improve perception additively.
  ACE is the commercially available, reference sound processing strategy.
  Cochlear Device Interface (CDI) Tool: For all strategies, programming will be performed using a research version of Custom Sound and the investigational software: CDI Tool.
Arm/Group | All Participants
Number analyzed (Participants) | 8
Percentage of words repeated correctly
  ACE Strategy | 51 (14.97)
  SPACE Strategy | 51.25 (10.95)
  OPAL-SPACE Strategy | 48.50 (14.45)

ADVERSE EVENTS:
Time Frame: 6 weeks (Time from treatment assignment to End of Study visit)
Groups:
- All Participants: Advanced Combination Encoder (ACE) sound processing strategy (reference strategy), Spread Precompensation Advanced Combination Encoder (SPACE), and Optimised Pitch and Language strategy-SPACE (OPAL-SPACE; combined OPAL and SPACE strategy) were evaluated in adult cochlear implant recipients. All strategies were programmed using a research version of Custom Sound and the investigational software: Cochlear Device Interface Tool (CDI Tool).
Arm/Group | All Participants
All-Cause Mortality (participants affected / at risk) | 0/8
Serious Adverse Events (participants affected / at risk) | 0/8
Other Adverse Events (participants affected / at risk) | 0/8

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-06-03): https://cdn.clinicaltrials.gov/large-docs/28/NCT05476328/Prot_SAP_000.pdf